CLINICAL TRIAL: NCT05073328
Title: Burden of Care of Long COVID Patients After Hospital Discharge
Acronym: BLOC
Status: Completed | Type: Observational
Sponsor: Mikhail Dziadzko, MD, PhD (Other)
Collaborators: PELyon (Unknown)
Responsible Party: Sponsor-Investigator, Mikhail Dziadzko, MD, PhD, Principal Investigator, Hôpital de la Croix-Rousse
Organization: Hôpital de la Croix-Rousse (Other)
Other Study IDs: BLOC-HCL/PELyon
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; COVID Long
Keywords: COVID-19; Long COVID; Long-haul COVID-19; post-COVID-19 pain; chronic pain; burden of care; care consomption; national database
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 patients: COVID-19 patients discharged from all French hospitals from 01 February to 30 June 2020
  Interventions: Other: COVID-19 required hospitalisation
- sub group The "long COVID" patients: this cohort will include patients with at least 4 weeks of claims and specific health care use after hospital admission from the initial cohort (COVID-19 patients)
  According to the Haute Autorité de Santé (HAS), the most frequent symptoms in the context of long COVID are the following :
  * Major fatigue
  * Dyspnoea, cough
  * Chest pain, often tightness type, palpitations
  * Problems with concentration and memory, lack of words
  * Headache, paraesthesia, burning sensation
  * Disorders of smell, taste, tinnitus, dizziness, odynophagia
  * Muscle, tendon or joint pain
  * Sleep disorders (especially insomnia)
  * Irritability, anxiety
  * Abdominal pain, nausea, diarrhea, decrease or loss of appetite
  * Pruritus, urticaria, pseudo-frostbite
  * Fever, chills
  Interventions: Other: COVID-19 required hospitalisation
- sub group "non long COVID" patients: all other patients from the initial cohort (COVID-19 patients )
  Interventions: Other: COVID-19 required hospitalisation

INTERVENTIONS:
Other: COVID-19 required hospitalisation — Patients who contracted a COVID19 required hospitalisation

SUMMARY:
Since March 2020, 3.5 million people have been infected with SARS-COV2 in France, and about 250 000 patients have been hospitalized and successfully discharged.

In a majority of cases, the evolution of the disease is favourable, but both hospitalized or patients with a mild form of the disease may present so called "Long-COVID" syndrome - a patient-created term which describes the effects of COVID-19 that continue for weeks or months beyond the initial symptoms. There is thus an urgent need to evaluate the long-term medical resource utilisation (MRU) and health care burden incurred by patients with Long-COVID, as well as risk factors for Long-COVID.

We will use the SNDS database to extract and analyze the data relevant to the project objectives. Indeed, the SNDS database is the French NHS database providing individual anonymous information of primary and secondary care linked at individual level (data from PMSI, the French DRG-based medical information system). It currently covers more than 98% of the French population.

For the first time, our study will provide an estimation of MRU and associated costs of hospitalized COVID-19 patients. It will also provide an estimation of the rate of long COVID forms developed by hospitalized COVID patients, as well as detailed MRU and costs incurred by long COVID patients compared to patients with non-long COVID-19.

DETAILED DESCRIPTION:
Since March 2020, 3.5 million people have been infected with SARS-COV2 in France, and about 250 000 patients have been hospitalized and successfully discharged . Currently, the French epidemiological situation shows a stable and high level of new cases of COVID-19 (around 20 000 per day) and associated hospitalizations (around 9 000 per week).

COVID19 may present mild or severe forms, the latter possibly requiring conventional (20%) or intensive care unit (ICU) hospitalization (5%). In most cases, the evolution of the disease is favorable, but both hospitalized or patients with a mild form of the disease may present so called "Long-COVID" syndrome - a patient-created term which describes the effects of COVID-19 that continue for weeks or months beyond the initial symptoms. Persistent symptoms have been described in 5 to 36% of the patients, i.e. symptoms persisting for 4 weeks or more after the onset of the disease. There is growing evidence of the post-COVID-19 chronic syndrome as a postinfectious entity, including but not limited to a range of symptoms ranging from cough and shortness of breath, to fatigue, headache, palpitations, chest pain, joint pain, physical limitations, depression, and insomnia, persisting for longer than two months. This post-COVID chronic syndrome is often called "long COVID". As it is more and more described since the start of the pandemic, the French national health agency (Haute Autorité de Santé, HAS) has recently published specific recommendations for the management of patients presenting long COVID forms.

Although the evidence is still scarce, patients who have been hospitalized for COVID19 may be at higher risk of presenting long COVID. Consequently, they may require more healthcare resource use. As they are easy to identify through administrative databases, we propose to focus on hospitalized and discharged COVID-19 patients with persisting symptoms, in order to investigate their healthcare resource use and corresponding costs, and to compared them to patients not presenting the long COVID form of the disease.

The objectives of this study are:

1. to assess "long-COVID" patients' health care burden (costs) and resource use and to compare them to COVID patients not developing the long form of the disease
2. to identify predictive variables for the development of "long-COVID",
3. to investigate whether different patterns of long-COVID healthcare consumption may be identified.

This will be performed using the Système National des Données de Santé (SNDS) French medico-administrative database.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Patients hospitalized between February 1st and June 30st 2020 for COVID-19 as the main diagnosis, using the following ICD-10 discharge codes: U07.10, U07.11, U07.14, U07.15
* Patients alive at the date of discharge

Exclusion Criteria:

* not affiliated to the French Social Security
* not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COVID-19 patients discharged from all French hospitals from 01 February to 30 June 2020
Sampling Method: Non-Probability Sample
Enrollment: 68822 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
MRU (medical resource use ) | 6 months following the discharge date
  The primary outcome will be the description of MRU and related costs during the 6 months following the discharge date, i.e.:
  * medications,
  * medical, including chronic pain structure consultation/admission,
  * emergency room visits
  * paramedical visits (e.g. nurse visits, physiotherapist, psychologist)
  * specific therapies including pain management,
  * medical procedures, biological acts
  * new hospitalizations (for any reason),
  * sick leaves,
  * transportation

SECONDARY OUTCOMES:
Predictive variables for "long-COVID" | up to 1 year before the hospitalisation date
  identified risk factors for developing long-COVID
Patterns of long-COVID healthcare consumption | 6 months following the discharge date
  typologies of consumption (cluster analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail DZIADZKO, MD, PhD, Principal Investigator — Hospices Civils de Lyon; Frederic Aubrun, MD, PhD, Principal Investigator — Hospices Civils de Lyon; Eric VAN-GANSE, MD, PhD, Principal Investigator — Hospices Civils de Lyon; Pierre ALBALADEJO, MD, PhD, Study Chair — CHU Grenoble Alpes; Florence ADER, MD, PhD, Study Chair — Hospices Civils de Lyon; Valeria MARTINEZ, MD, PhD, Study Chair — Hôpital Raymond-Poincaré - APHP; Claire MARANT-MICALLEF, PharmD, MPH, Study Director — PELyon; Manon BELHASSEN, MD, PhD, Study Director — PELyon; Fabrice HERITIER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital de la Croix Rousse - Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No
individual participant data are protected by the French legislation and are not shared

REFERENCES:
- [Derived] Dziadzko M, Belhassen M, Van Ganse E, Heritier F, Berard M, Marant-Micallef C, Aubrun F. Health Care Resource Use and Total Mortality After Hospital Admission for Severe COVID-19 Infections During the Initial Pandemic Wave in France: Descriptive Study. JMIR Public Health Surveill. 2024 Sep 11;10:e56398. doi: 10.2196/56398. PMID 39259961